CLINICAL TRIAL: NCT02085694
Title: A Pilot Study on the Efficacy of Lactobacillus Brevis CD2 Lozenges in Preventing Oral Mucositis by High-dose Chemotherapy With Autologous Hematopoietic Stem Cell Transplantation
Brief Title: Lactobacillus Brevis CD2 Preventing Oral Mucositis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, sabrina giammarco, MD, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 001/14
Record Dates: First submitted 2014-03-06; First posted 2014-03-13 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Mucositis
MeSH Terms: conditions — Mucositis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lactobacillus brevis CD2 lozenges (Experimental)
  Interventions: Drug: Lactobacillus brevis CD2

INTERVENTIONS:
Drug: Lactobacillus brevis CD2

SUMMARY:
A pilot study on efficacy of Lactobacillus CD2 lozenges in preventing oral mucositis (OM) by high-dose chemotherapy with autologous hematopoietic stem cell transplantation. To test whether the probiotic Lactobacillus brevis CD2 lozenges can reduce the incidence and severity of high-dose chemotherapy conditioning regimen induced OM in patients undergoing HSCT.

Clinical activity will be defined as reduction in the incidence of chemotherapy induced OM in the patients undergoing HSCT.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Karnofsky Performance Score ≥ 70%.
* Confirmed histological diagnosis of multiple myeloma for which HSCT is as approved modality of therapy
* Patients eligible to receive high-dose chemotherapy as part of conditioning regimen
* Concomitant co morbid condition if present, controlled by ongoing treatments (e.g. hypertension, diabetes and so on)
* Serum creatinine < 1.8mg/dl
* Total bilirubin < 2mg/dl
* Liver enzymes within three times of normal limit
* Expected survival > 6 months.

Exclusion Criteria:

* Pregnant women and lactating mothers
* Patients with history of HIV infection
* Patients who have taken any other investigational product in last 4 weeks
* Patients having untreated symptomatic dental infection
* Patients with WHO Grade 3 or 4 oral Mucositis
* Other serious concurrent illness
* Inconclusive hematological diagnosis
* Patients with signs and symptoms of systemic infections
* Patient's/guardian's refusal to sign informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-11 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
COMMON TERMINOLOGY CRITERIA FOR ADVERSE EVENTS v4.03 (CTCAE) for evaluation of change in oral mucositis | days -14;-7; 0;+7;+14;+21

SECONDARY OUTCOMES:
COMMON TERMINOLOGY CRITERIA FOR ADVERSE EVENTS v4.03 (CTCAE) to determine the incidence of Grade I and II OM | days -14;-7; 0; +7;+14; +21

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Universitario "A. GEMELLI", Rome, Rome, Italy